CLINICAL TRIAL: NCT00565942
Title: Exploring Integrative Medicine for Back and Neck Pain - A Pragmatic Randomized Clinical Pilot Trial
Brief Title: Exploring Integrative Medicine in Swedish Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ekhagastiftelsen (Other); Insamlingsstiftelsen för forskning om manuella terapier (Unknown); Primary care units at Bagarmossen, Skarpnäck, Dalen and Björkhagen (Unknown); Svensk förening för vetenskaplig homeopati (Unknown); HRQL gruppen, Göteborgs universitet (Unknown)
Responsible Party: Principal Investigator, Torkel Falkenberg, Researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM in Swedish primary care
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Back or Neck Pain of at Least 2 Weeks Duration
Keywords: Integrative medicine; Primary care; Swedish massage therapy; Manual therapy; Naprapathy; Shiatsu; Acupuncture; Qigong; Pragmatic ranomized controlled pilot trial; Health services research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Treatment as usual coordinated by general practitioners in primary care.
  Interventions: Procedure: Usual care
- Integrative care (Active Comparator): Selected complementary therapies (Swedish massage therapy, manual therapy/naprapathy, shiatsu, acupuncture and qigong) added to usual care.
  Interventions: Procedure: Integrative care

INTERVENTIONS:
Procedure: Integrative care — In short, integrative care was up to 10 complementary therapy treatments delivered to the patient in addition to the usual care over an intervention period of up to 12 weeks. The integrative care was provided by a multidisciplinary team coordinated by a gate keeping general practitioner with clinical knowledge and experience of CTs and senior licensed/certified CT providers representing Swedish massage therapy, manual therapy/naprapathy, shiatsu, acupuncture and qigong.
  Arms: Integrative care
Procedure: Usual care — The usual care treatment was coordinated by the patient's general practitioner and complied with the clinical practice routines at the participating primary care units. Conventional procedures included but were not exclusive to advice, prescription of drugs, sick leave and physiotherapy/physical therapy. There were no constraints to the provided usual care as the study aimed to pragmatically reflect the general practitioners' standard care and treatment as usual.
  Arms: Usual care

SUMMARY:
Research over the last years have reported an increased popularity of complementary therapies (CTs) and an integration of CTs into mainstream medical settings, health care organizations and insurance plans. These trends may present both new challenges and new opportunities for health care provision. In Sweden and elsewhere, major challenges include the great variety and quality of CT provision within health care and a lack of national and international recommendations of how integrations of CTs with conventional care should be modelled, i.e. lack of conceptual models for delivering integrative medicine (IM). This may partly be a result of a scarce evidence base in support of IM provision within public health care services, e.g. lack of IM compared to usual care in randomised clinical trials. It remains largely unknown whether comprehensive models of IM are clinically or cost effectively different from conventional care provision.

Back and neck pain are costly, conventionally managed in primary care and two of the most common conditions treated by CTs. We have developed a comprehensive collaborative consensus model for IM adapted to Swedish primary care. The aim of this pilot study was to explore the feasibility of a pragmatic randomised clinical trial to investigate the effectiveness of the IM model versus conventional primary care in the management of patients with non-specific back/neck pain.

DETAILED DESCRIPTION:
Study objectives included the exploration of recruitment and retention rates, patient and care characteristics, clinical differences and effect sizes between groups, selected outcome measures and power calculations to inform the basis of a full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Back/neck pain with or without headache for at least two weeks and at least three times per week
* Resident of Stockholm County
* Literate in Swedish
* Willing and able to comply with study requirements

Exclusion Criteria:

* Specific pathology and severe causes of back/neck pain such as malignant disease, vertebral fractures and severe or progressive neurological symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Days with pain | Change from baseline to follow-up after 16 weeks
  Number of days with pain over the last two weeks (0-14 days)
Physical functioning | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Role physical | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Bodily pain | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
General health | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Vitality | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Social functioning | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Role emotional | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Mental health | Change from baseline to follow-up after 16 weeks
  SF-36 domain 0-100 (higher score better)
Disability | Change from baseline to follow-up after 16 weeks
  Numerical rating scale 0-10 (higher score worse)
Stress | Change from baseline to follow-up after 16 weeks
  Numerical rating scale 0-10 (higher score worse)
Well-being | Change from baseline to follow-up after 16 weeks
  Numerical rating scale 0-10 (higher score better)
Use of prescription analgesics | Change from baseline to follow-up after 16 weeks
  Use of prescription analgesics during the last two weeks (yes/no)
Use of non-prescription analgesics | Change from baseline to follow-up after 16 weeks
  Use of non-prescription analgesics during the last two weeks (yes/no)
Use of conventional care | Change from baseline to follow-up after 16 weeks
  Use of conventional care during the last two weeks (yes/no)
Use of complementary care | Change from baseline to follow-up after 16 weeks
  Use of complementary care during the last two weeks (yes/no)

OTHER OUTCOMES:
Recruitment of patients | At baseline
  Number of included patients at baseline
Retention of patients | After 16 weeks
  Number of patients completing follow-up after 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Torkel Falkenberg, PhD, Principal Investigator — Karolinska Institutet, Department of Neurobiology, Care Sciences and Society, Division of Nursing
Locations (1):
- Karolinska Institutet, Department of Neurobiology, Care Sciences and Society, Division of Nursing, Huddinge, Sweden

REFERENCES:
- [Background] Sundberg T, Halpin J, Warenmark A, Falkenberg T. Towards a model for integrative medicine in Swedish primary care. BMC Health Serv Res. 2007 Jul 10;7:107. doi: 10.1186/1472-6963-7-107. PMID 17623105
- [Result] Sundberg T, Petzold M, Wandell P, Ryden A, Falkenberg T. Exploring integrative medicine for back and neck pain - a pragmatic randomised clinical pilot trial. BMC Complement Altern Med. 2009 Sep 7;9:33. doi: 10.1186/1472-6882-9-33. PMID 19735542